CLINICAL TRIAL: NCT02404727
Title: Evaluation of Cemented and Cementless Fixation of Dual-mobility Hip Prosthesis in Elderly Patients With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Holstebro Hospital
Record Dates: First submitted 2015-01-21; First posted 2015-03-31 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2014-12

CONDITIONS: Osteoarthritis, Hip; Arthropathy of Hip
Keywords: Osteoarthritis, Hip; acetabular fixation; dual mobility cup; Radiostereometric Analysis; Dual-Energy Radiographic Absorptiometry; Accelerometry; total hip arthroplasty; intra-prosthetic dislocation
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cup fixation cemented (Active Comparator): 30 of the 60 patients will be randomized to cemented cup fixation
  Interventions: Procedure: cup fixation; Device: Avantage® Cup
- cup fixation cementless (Active Comparator): 30 of the 60 patients will be randomized to cementless cup fixation
  Interventions: Procedure: cup fixation; Device: Avantage® Cup

INTERVENTIONS:
Procedure: cup fixation — All patients will preoperatively, 3 months, 1 year, 2 year and 5 year have the hip DXA scanned, answer PROM, X-ray for RSA analysis and wear measurements, and wear accelerometry chip 14 days prior each outward clinic visit for movement analysis.
Device: Avantage® Cup

SUMMARY:
The aim of this project is to investigate prosthesis fixation in the bone, respectively cemented and uncemented operation method of Avantage® dual-mobility acetabular cup in elderly patients, wear of the plastic in dual-mobility hip prosthesis and evaluate the clinical function, patient satisfaction and possible complications.

Patients included in this study suffer from osteoarthritis of the hip.

DETAILED DESCRIPTION:
The Elderly Hip Patient The proportion of elderly in the Danish population is increasing and their and functional level is generally good, despite other health problems, which intensifies the demand for a primary definitive (one-stage) and safe surgical treatment in case of osteoarthritis or fragility low-energy displaced femoral neck fracture. Total hip arthroplasty (THA) is one of the most successful procedures in modern orthopaedic surgery to achieve pain relief and restore normal walking ability in a preoperative painful and stiff hip joint.

Bone Quality and THA surgical technique Osteoporosis (brittle bones) is defined as a chronic systemic skeletal disease characterized by low bone mineral density (osteopenia) and microarchitecture changes in the trabecular bone structure resulting in reduced strength and therefore increased risk of fractures. Among Danish women over 65 years of age, the prevalence of osteoporosis is 40-60%, and the prevalence among men is increasing. Much effort is put into secondary fracture prophylaxis such as vitamin D and calcium as well as medical bone anti-resorptive treatment (i.e. bisphosphonates).

When the bone is weak/osteoporotic there is a general but undocumented recommendation of cemented over uncemented THA fixation. It has been shown that uncemented hip stems migrate more than cemented components in osteopenic and osteoporotic bone wherefore cemented stem fixation is recommended. However, Danish hip surgeons favour uncemented fixation even in the fragile and osteoporotic elderly because it reduces the surgical time, minimizes the risk of intraoperative cement disease/fat embolism and dead, and makes revision surgery in case of infection or peri-prosthetic fracture easier to re-operate. In 2012, 7364 acetabular cups were inserted uncemented versus 1015 uncemented - for all indications for THA in Denmark. Reoperation of the same hips within 2 years after primary THA due to new femoral neck fracture or complications following treatment of proximal femoral fracture was 4.7 %. There is clinical conviction that cemented cups are easier to place in the correct inclination and anteversion position. However, due to the posterior-lateral overhang of dual mobility cups the postero-lateral edge-cementation is likely to be insufficient leading to micromotion and aseptic loosening. In the clinical experience this is a lesser risk with cementless cups. Compared to other Nordic countries, Denmark has the lowest incidence of aseptic cup loosening of 34.8% and respectively 47.3% and 50.4% for Norway and Sweden. The reason for revision due to dislocation is 33.5% in Denmark compared to Norway and Sweden, respectively 23.8% and 23.4% and may be related to an overall difference in surgical approach (postero-lateral approach in Denmark but antero-lateral approach in Norway and Sweden). Approximately 96% are operated with posterior approach in Denmark whereas 23.8% and 60.3% were operated by posterior approach in Norway and Sweden, respectively.

Dual-mobility articulation concept In 1974 Professor Bousquet developed the dual-mobility (DM) hip articulation concept to reduce wear, restore near-normal motion-range in the hip joint, and at the same time increase hip prosthesis stability. The dual-mobility hip articulation design consist of a large non-fixed polyethylene liner sliding freely within the metal cup-shell which is fixed into the bone, and inside the mobile liner is a second articulation with a small femoral head. The dual-articulation of the prosthetic joint prevents impingement of the femoral neck on the acetabular rim of the implant. Studies have shown that dual-mobility hip prostheses have good survival rates and reduces dislocation rates both in patients with primary osteoarthritis of the hip and a lesser compliant patient group with displaced femoral neck fractures . Clinical expectations for the dual-mobility articulation concept for treatment of displaced medial FNF are good; however, there are only a few publications available and there are no studies of implant fixation / cup migration. It is important to study both the dislocation risk as well as the mechanical stability of the bony fixation since the advantage of a low dislocation rate would be meaningless if the cups were to loosen mechanically from the surrounding bone in the mid- or longer term.

Femoral Neck Fracture and THA THA may be used as the primary treatment option for displaced medial femoral neck fractures (FNF). Compared to screw osteosynthesis, THA results in a stable fracture treatment with less post-operative pain and faster mobilization after displaced medial FNF and with fewer complications. The most common complication to THA treatment in old and perhaps memory-impaired patients is dislocation instability. At the Regional Hospital Holstebro our results with the Saturne® Dual-Mobility THA in this patient group (n>500) during the last 7 years propose the risk of THA hip dislocation in high-risk patients to be below 5%. In 2012, 10,309 patients were admitted to Danish hospitals with femoral fractures. Approximately 600 of these hip fracture patients were treated with THA. Patients with hip fractures are very resource intensive and require approximative 2.2% of all hospital bed days in Denmark. Furthermore, these elderly, with an average age of 80 years and a high co-morbidity percentage also have a high mortality risk of approximately 10% within the first 30 days after FNF. The one-year mortality is 15-25%. Reoperations frequency depends on the fracture type and operative treatment, and varies from a few per cent after insertion of THA to 25% after osteosynthesis. Often it is the acute and chronic medical conditions that cause the elderly to low energy falls resulting in hip fracture, but it may also just be accidental and related to osteoporosis.

Radiostereometric Analysis (RSA) Mechanical loosening of the prosthesis may be suspected if the prosthesis migrates relative to underlying and adjacent bone. Therefore, there is now a consensus that the introduction of new prostheses and new operational methods of prosthesis insertion should be evaluated through migration studies before they can be recommended for use in general. Clinical studies have shown a high predictive power between early migration of joint prostheses and later prosthesis loosening and premature revision. Radiostereometric analysis (RSA) is a very accurate method for assessment of cup migration at precision levels 0.11 mm precision or better.

Dual Energy X-ray Absorptiometry (DXA) The clinical survival of joint prostheses depends on the quality of the surrounding bone and bone mineral density (BMD) is an important measure of bone strength and quality. The periprosthetic bone density can be measured with Dual Energy X-ray Absorptiometry (DXA), which is a precise method for measuring even small changes in BMD around hip prostheses. Patients are exposed to a very little dose of radiation with these studies and scanning only takes a few minutes. Typically, four to five scans are taken during a 2 to 5 year follow-up. For assessment of the bone surrounding the acetabular cup the 3 DeLee zones or the 4 Wilkinson Zones are often used, and Gruen zones are used for assesment around the stem.

Bone density is defined by a and in osteopenic bone the T-score is between <1.0 - > 2.5, whereas when osteoporotic the T-score is < 2.5 and severe osteoporosis < 4.0.

It is possible to register bone resorption around implants with DXA before resorption becomes visible on conventional x-ray films in the form of "radiolucent lines" (RLL). It is important to monitor remodelling in the periprosthetic bone because decreasing BMD may weaken the prosthetic fixation and lead to failure. It is known that BMD decreases initially after implant surgery and then stabilize after a periode of a few years.

Polywear The acetabular plastic component polyethylene (PE) wear particles stimulate a biologic response with production of various inflammatory mediators, which stimulate migration of leucocytes into tissues and activate collagen synthesis, and stimulate osteoclasts to resorb bone and contribute to osteolysis.

Reports have suggested that hydroxyapatite (HA) coated implants that are used in cementless hip replacements further contribute to inferior survival of medium- thickness spray-dried HA-coated cups with individual cases of excessive PE wear and premature cup failure.

The concept of the dual-mobility cup provides a theoretical question whether the double articulations leads to more wear and hence earlier revision, especially in younger more active patients.

It has previously been shown that a two-dimentional (2D) wear of the polyethylene of 0.1 mm / year may lead to osteolysis and loosening of the prosthetic components, which deteriorates prosthesis durability.

Wear of hip prostheses polyethylene can be accurately measured (0.09 mm) with software PolyWare 3D Pro Digital Version on digital clinical antero-posterior radiographs of the hip prosthesis.

Study design and methods Comparison of prosthesis migration of cemented versus uncemented dual-mobility cup fixation Objective: Investigate prosthesis migration and polyethylene wear of cemented and cementless Avantage® dual-mobility acetabular components (Biomet Inc.) in elderly patients and correlate migration measurements with radiological evaluation of implant placement/cementation quality, with bone quality at the time of surgery (osteoporotic/osteopenic/normal bone), and with functional outcome after two years. The migration pattern and magnitude will predict the likelihood of later aseptic loosening and revision.

Design:

Prospective randomized patient-blinded clinical trial.

Hypotheses:

1. More stable fixation of cemented compared with uncemented cups (initially and between 1-2 years).
2. Acceptable cement coverage at the postero-lateral acetabular rim in most (95%) of cases.
3. Low polyethylene wear-rate (<0.1mm/year after bedding-in during the first 3 months).
4. Similar periprosthetic pelvic bone loss (Wilkinson zones) irrespective of fixation method.
5. Low dislocation risk irrespective of fixation method (<1%).
6. Patient satisfaction >90% in general.

Patients:

The Avantage® cup is used for all elderly patients on our department including patients with displaced medial FNF and patients with primary osteoarthritis. It may also be used for revision surgery in case of dislocation complications. Acute patients with FNF are difficult to include in studies when some pre-study investigations are necessitated and further patients with FNF are difficult to inform (pain and morphine drugged) and it is difficult to give proper time to consider study participation and perhaps call for an assessor to help make the decision. A big drop out due to difficult circumstances about project-information and consent could be a serious selection bias and could also prolong the inclusion period seriously. Mortality in FNF patients is high and poses a risk of many patients lost to follow-up during a 5-year study period and therefore demands a high estimated sample size. Therefore this study applies only to elderly elective patients with osteoarthritis scheduled for elective THA. All patients >70 years of age with osteoarthritis of the hip, who are candidates for a total hip prosthesis, will be offered participation in the study. All patients will be operated by one of two experienced hip surgeons and they will follow the usual postoperative regime at Holstebro Regional Hospital (pain treatment, physiotherapy and full weight bearing, thromboembolic and antibiotic prophylaxis). All eligible patients will be registered, those who choose not to participate, will be asked for the reason of refusal, to be able to detect possible selection bias.

INFORMED CONSENT The first contact is made in the outpatient clinic of orthopaedic department of Regional Hospital Holstebro, where the patients will be seen by one of two orthopaedic surgeons experienced in total hip replacement surgery.

With the first contact, the patients will receive oral and written information about the study. During this contact it is possible for the patient to have an extra person along. If requested by the patient/needed for decision-making concerning study participation, we will offer second project information to the patient with the option to bring an assessor. Patients can decide to participate in the study up to a week before surgery, where they will come to the information day prior to surgery, which is a part of the normal fast-track program. There is an average waiting period between first contact and surgery of 4 weeks, which means that patients have 3 weeks to decide. Written informed consent will be obtained before commencement of data collection, at the latest on the information day prior to surgery. When the consent form is signed DXA scanning and filling out questionnaires will commence, and post-operative stereoradiographs and DXA scans will be booked.

Method:

All patients will be DXA scanned pre-operatively for measurements of general bone mineral density and classification in a) normal bone, b) osteopenia) or c) osteoporosis. Patients with a T-score above -2.5 (normal bone and osteopenic bone) will be grouped and patients with a T-score at or below -2.5 and at or above - 4.0 will be grouped (osteoporosis). Patients will be stratified to the two treatment modalities (cemented acetabular cup fixation and cementless acetabular cup fixation) according to this dichotomy on T-score. Patients with a new diagnosis of osteoporosis will be referred to their own general practitioner concerning blood work and initiation of anti-resorptive treatment. On going medical treatment for osteoporosis will be recorded. After stratification according to T-score, patients are randomized during surgery with a cemented or cementless Avantage® dual-mobilty Cup (Biomet Inc.) and patients will be blinded with respect to implant fixation method. The Avantage® Cup can be inserted both cemented and uncemented where the cementless are HA coated and cemented cups are fully polished. The liner is gamma irradiated to induce a high level of crosslinking and Vitamin E is infused into the highly crosslinked polyethylene. A 28-mm chrome-cobalt femoral head will be used in all cases. The femoral stems will be similar in all patients (cemented Exeter stems, Stryker® Inc.) and Palacos® bone cement (Heraeus Medical inc.) will be used. During surgery 1mm tantalum beads are inserted in the bone surrounding the prosthetic components (both the femur and the cup) allowing for post-operative migration measurements with RSA.

Postoperative, 3 months, 1 year, 2 years and 5 years after surgery the patients are followed with:

* Stereo radiographs (cup migration and polyethylene wear).
* Standard radiographs (evaluation of cup position (PolyWare software) and evaluation of cementation quality)
* DXA scan at follow-up to measure changes in the peri prosthetic bone density (Wilkinson Zones in the acetabulum and Gruen Zones around the stem).
* Collection of PROM (Osteoporosis risk assessment, Oxford Hip Score,EuroQol-5D (EQ-5D), Harris Hip Score, VAS score at rest and activity).
* Activity measurement with an accelerometer 2 weeks test prior to each control.

Power and data analysis: The proximal cup migration was used as the primary effect variable in the pre-study power analysis based on a pilot study including both cemented and cementless Avantage DM cups. Sample size calculation using two-sample mean test for a minimal relevant difference of 0.2mm with a mean cup migration of 0.1mm and a standard deviation of 0.2 (pilot study), power of 0.90, and 5% risk of type-1 error, 23 patients were needed in each group. To compensate for potential dropouts, we decided to include 30 hips in each treatment arm. Secondary endpoints are polyethylene wear, activity, complications, and functional outcome by clinical examination (HHS) and PROM (OHS, EQ5D). All of the applied methodologies are available, accessible and validated at Holstebro Regional Hospital.

The Helsinki II agreement will be followed. The study plan will be registered at clinicaltrails.gov. Application for permission for a database will be submitted to the Data Protection Agency of the region Midtjylland and data will be stored in accordance with applicable law.

Ethics and (dis) advantages for the patient There are only a few publications available on implant fixation in elderly patients and currently only for fixation of the stem in patients with normal bone or osteoporotic bone. There are no RSA studies available on the Avantage® cup even though it is the standard cup in most Danish Orthopaedic Departments and one of the cups available in the Middle Region Implant Supply. The Avantage® cup is available in a similar design for cemented and cementless fixation principle. The dual-mobility concept is well proven in different implant brands over 35 years with good results on revision and dislocation (both very low) but no RSA studies on fixation are available. The current study may therefore add important and new knowledge to the literature. It is important to study both the dislocation risk as well as the mechanical stability of the bony fixation since the advantage of a low dislocation rate would be meaningless if the cups were to loosen mechanically from the surrounding bone in the mid- or longer term.

The study will reveal insight into whether the cemented or the cementless fixation principle is better for elderly patients and if there is a difference based on systemic and periprosthetic bone mineral density. Furthermore compiled prosthesis migration with the bone quality, accelerometer tests, and the incidence of complications that could contribute to the improvement of hip prosthesis surgery to such an extent that clearly outweighs the side effects associated with the study.

The study will be performed using the fast-track program of the department, ensuring the same length of stay for both groups, and no additional admission days are added as compared to other patients who undergo hip prosthesis surgery. Patients have minimal increased radiation dose compared to the usual control regime after hip replacement surgery. Written and informed consent is required. The local research ethics committee must approve the study before initiation.

Measurements were taken for the radiation dose, which shows that the stereo x-ray of the hip provides a very low radiation dose of 0.15 mSv.. DXA measurements of the femur or spine (osteoporosis control) produce an effective dose equivalent to 292 millisievert (milliSv) and a scan around the hip implants produce an effective dose of 146 milliSv (info from General Electric (GE) scanner manufacturer). A conventional radiograph of the hip provides a dose of 0.85 milliSv. Patients, who undergo hip prosthesis surgery outside the protocol in our hospital unit, have one conventional radiograph after surgery and, as of recently, no clinical or radiographic later follow-up due to necessary cuts on budget-costs. Patients in this study have one conventional radiograph post-operatively and one conventional x-ray at 2 years and 5 years follow-up. In total the project patients are subjected to an additional radiation dose of 2 conventional radiographs (1.7 mSv), 1 osteoporosis assessment (0.03 mSv), seven times periprosthetic DXA scans including double measurements (0.1 mSv) and six times the stereo radiography including double measurements (0.9 mSv). Patients included in this study get exposed to an additional radiation dose of 2.73 mSv. This corresponds to approximately 3 conventional radiographs of the hip, and it provides an additional risk of fatal cancer of 0.01%. This places the subjects in group IIb., where the overall risk of the irradiated individual is 1 to 10,000.

No financial support/compensation will be offered to patients for study participation. Regarding compensation and remuneration after death or injury of a project participant reference is to the national patient insurance program.

Publication of results The project is part of a Doctor of Philosophy (Ph.D.) project concerning treatment of dislocated Garden I and II femoral neck fracture with a dual-mobility arthroplasty concept. The Ph.D. protocol has been approved for enrollment at Aarhus University Hospital during spring/summer 2014. All results, both positive and negative as well as inconclusive, will be sought published in international scientific peer-reviewed journals as well as presented on national and international scientific conferences. The Vancouver rules for authorship will be followed. There is a mutual agreement that Steffan Tábori Jensen will write the manuscript as the first author.

Previous RSA and research at Holstebro Regional Hospital The Orthopaedic Research Unit, Regional Hospital Holstebro, has the needed technical research staff and academic research expertise, the required experience and software/equipment, including server capacity and software, to complete the study. Several articles in this area have been published emanating from the department and its associates.

ELIGIBILITY:
Inclusion Criteria:

1. Both men and women with osteoarthritis of the hip joint.
2. Patients with adequate bone quality for insertion of a cementless acetabular component.
3. Age 70 years and above, capable and empowered.
4. Informed written consent.
5. The patient may only participate with one hip.

Exclusion Criteria:

1. Patients with severe nerve, muscle and vascular disease in the lower extremities
2. Patients that during surgery are assessed not suitable for treatment with cementless hip prosthesis.
3. Patients with severe osteoporosis (T-score < 4.0) as assessed by DXA scan before surgery..
4. Patients with previous hip fractures.
5. Patients who have previously undergone correction of bone malalignment of the hip or other major hip surgery.
6. Patients in need of a different stem that the Exeter stem (Stryker inc.).
7. Patients with metabolic disease of the bone or arthritis.
8. Patients who needing treatment with corticosteroids in tablet form (> 3 months / year).
9. Patients with metastatic cancer and / or radiation therapy and / or chemotherapy.
10. Patients without Danish citizenship / patients who do not speak and understand Danish.
11. Senile dementia.
12. Alcoholism (more than 21 drinks / week for men and more than 14 drinks / week for women).
13. Severe psychiatric illness.
14. Severe systemic disease affecting gait and mobilization (e.g. Parkinson's disease or hemiplegia). Very poor dental status (risk of infection).

Exclusion criteria after operation

1. Senile dementia / lost impartiality
2. Metastatic cancer and treatment with radiation and / or chemotherapy
3. Massive new systemic sickness (e.g. Hemiparesis or Mb. Parkinson).
4. Infection that leads to replacement of the acetabular component.
5. Fracture in relation to the prosthesis.
6. Immobilization in longer (> 3 month) periods (e.g. in relation to lower leg fracture or sickness)
7. Replacement of the acetabular component during the period of the project (e.g. due to loosening of the prosthesis without infection)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Cup migration, measured by Radiostereometric Analysis | 5 years
  cup migration in the cemented and cementless cups are measures with Radiostereometric Analysis.
  The primary endpoint was proximal cup migration (y-axis) at the 2-year follow-up.

SECONDARY OUTCOMES:
Polyethylene wear, measured by Radiostereometric Analysis | 5 years
  measurement af the plastic (polyethylene) are measured with Radiostereometric Analysis.
Bone mineral density, measured by dual energy X-ray Absorption (DXA) scans | 5 years
  Dual energy X-ray Absorption (DXA) scans are made to measure to bone mineral density around the prosthesis.
PROMS | 5 years
  Patient Reported Outcome Measures (PROM) are collected continuously
Physical activity monitoring and classification, motion analysis. | 5 years
  3-axis accelerometer. Monitor human movements continuously to determine pre and postoperatively movements, mobility and activity for the assessment of functional ability.
  The Activity (AX3) device is securely fastened to the patients hip two weeks preoperatively and again two weeks prior to each outward clinic visit at 3 months, 1 yr, 2 yr and 5 yr.

CONTACTS AND LOCATIONS:
Overall Officials: Torben B. Hansen, Ph.D., Professor, Study Director — Department of Orthopaedic Surgery, Hospital Unit West, Denmark
Locations (1):
- University Clinic of Hand, Hip and Knee Surgery, Holstebro Hospital, Holstebro, Denmark